CLINICAL TRIAL: NCT00898014
Title: Study Evaluating the Prognostic and Predictive Value of Response to First-Line Chemotherapy by Detection of Circulating Tumor Cells (CTC) in Patients With Metastatic Breast Cancer
Brief Title: Blood Levels of Tumor Cells in Predicting Response in Patients Receiving First-Line Chemotherapy for Stage IV Breast Cancer
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000574195; CLCC-IC-2006-04; INCA-RECF0474
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — In Situ Hybridization, Fluorescence; Immunologic Techniques

INTERVENTIONS:
Genetic: fluorescence in situ hybridization
Other: immunologic technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Measuring blood levels of tumor cells in patients with breast cancer may help doctors predict how patients will respond to treatment.

PURPOSE: This laboratory study is looking at blood levels of tumor cells in predicting response in patients receiving first-line chemotherapy for stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Predict the overall and progression-free survival of patients with stage IV breast cancer by measuring the rate of circulating tumor cells (CTC) before the second course of chemotherapy.

Secondary

* Predict overall and progression-free survival of these patients by measuring the rate of CTC before the start of chemotherapy, at the first tumor evaluation, and after 2-3 courses of chemotherapy.
* Correlate the detection of CTC with tumor markers, clinical response, and radiological response.
* Study the changing status of HER-2 in CTC in patients receiving trastuzmab (Herceptin®).

OUTLINE: This is a multicenter study.

Blood samples are collected at baseline, before the second course of chemotherapy, before the third or fourth course of chemotherapy, and when progressive disease is diagnosed (before second-line treatment is initiated). Circulating tumor cells from the blood samples are examined by immunofluorescence.

Patients are followed periodically for up to 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage IV breast cancer
* Measurable or evaluable disease
* Scheduled to receive first-line chemotherapy with or without trastuzumab (Herceptin®), depending on HER-2 status
* Histologic block available for confirming pathologic diagnosis and measuring HER-2 status via FISH

PATIENT CHARACTERISTICS:

* Life expectancy > 3 months
* No other cancer in the past 5 years except for basal cell skin cancer or epithelial in situ cancer of the cervix
* No geographic, social, or psychiatric reasons that would make treatment impossible

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Correlation of circulating tumor cells (CTC) with overall survival
Correlation of CTC with progression-free survival

SECONDARY OUTCOMES:
Correlation of circulating tumor cells with tumor markers, clinical response, and radiological response
Change in HER-2 status in patients receiving trastuzumab (Herceptin®)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Pierga, MD, PhD, Study Chair — Institut Curie
Locations (1):
- Institut Curie Hopital, Paris, France